CLINICAL TRIAL: NCT01703910
Title: Phase II Individualized Therapies Selection Study for Patients With Metastatic Colorectal Carcinoma According to the Genomic Expression Profile in Tumor Samples.
Brief Title: Study of Individualized Therapies Selection for Patients With Metastatic Colorectal Carcinoma According to the Therapeutic
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centro Nacional de Investigaciones Oncologicas CARLOS III (Other)
Collaborators: Hospital Universitario de Fuenlabrada (Other); Grupo Hospital de Madrid (Other); Apices Soluciones S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CNIO-GI-01-2012
Record Dates: First submitted 2012-10-08; First posted 2012-10-11 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-10

CONDITIONS: Adenocarcinoma of Colon; Adenocarcinoma of Rectum; Metastatic Disease
Keywords: Genomic expression profile in tumor samples; Adult patients; metastatic disease status and progression after two lines of systemic therapy
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Neoplasm Metastasis | interventions — Capecitabine; Cisplatin; Cetuximab; Doxorubicin; Fluorouracil; Gemcitabine; Irinotecan; Topotecan; Mitomycin; Oxaliplatin; Paclitaxel; Docetaxel; Pemetrexed; raltitrexed; Sorafenib; Erlotinib Hydrochloride; Vinorelbine; Dasatinib; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Active Comparator): Control treatment and will be treated with any of the schemes used in the study according to the discretion of the physician.
  Interventions: Drug: Arm A chemotherapy
- Arm B (Experimental): Treatment guided by the gene expression profiles obtained from the CTC
  Interventions: Drug: arm B chemotherapy

INTERVENTIONS:
Drug: Arm A chemotherapy
  Other Names: Capecitabine; Cisplatin; Cetuximab; Doxorubicin; Fluorouracil; Gemcitabine; Irinotecan; Topotecan; Mitomycin C; Oxaliplatin; Paclitaxel; Docetaxel; Pemetrexed; Raltitrexed; Sorafenib; Erlotinib; Vinorelbine; Dasatinib; Etoposide
  Arms: Arm A
Drug: arm B chemotherapy
  Other Names: Capecitabine; Cisplatin; Cetuximab; Doxorubicin; Fluorouracil; Gemcitabine; Irinotecan; Topotecan; Mitomycin C; Oxaliplatin; Paclitaxel; Docetaxel; Pemetrexed; Raltitrexed; Sorafenib; Erlotinib; Vinorelbine; Dasatinib; Etoposide
  Arms: Arm B

SUMMARY:
The purpose of this study is to assess the feasibility of selecting personalized therapies for colon cancer patients who have failed standard treatments, using a new methodology based on the determination of a profile of chemosensitivity by comprehensive genetic expression analysis from tumor samples.

DETAILED DESCRIPTION:
It is a prospective, randomized study in patients with metastatic colorectal carcinoma progressing after two lines of prior therapy. Patients will be randomized (1:1) to receive chemotherapy as determined by its oncologist or treatment according to chemosensitivity profile obtained. For obtaining the profile a histological tumor sample and a sample of venous blood in a tube with heparin standard are necessary . This latter sample will be processed to isolate circulating tumor cells by cell adhesion with matrix coated glass spheres. The RNA from these circulating tumor cells as well as from tumor cells of tumor biopsies from the same patients will be extracted by a standard procedure for extracting RNA for genetic expression analysis. Based on the analysis performed on tumor biopsy is generated a ranked list of potentially more effective treatments in every case

ELIGIBILITY:
Inclusion Criteria:

* Histological examination showed of metastatic colon carcinoma.
* Patients more than 18 years.
* Measurable disease according to RECIST 1.1 criteriso
* Life expectancymore than 3 months according to the criteria of the investigator.
* Goodoverall condition determined by the ECOG scale (score 0-1)
* Candidate for systemic treatment based on the profile of sensibility to drugs determined by genetic analysis of the tumor sample. Patients should have received at least two lines of standard treatment, including therapies antiEGFR in cases of tumors with Kras oncogene B-Raf and native (non-mutated).
* Availability of tumor tissue or potential for tumor biopsy correlation allowing the RNA expression profile with that obtained from the peripheral blood CTCs.
* Adequate hematologic function: ANCmore than 1.5 x 103 / L, platelet count absolute more than 100 x 109 / L, normal values of INR and PTT.
* Adequate liver function: total serum bilirubin no more than 2 mg / dL, ALT and AST no more than 3 times the upper limit established by the laboratory (LSR) or no more than 5 LSR in patients with liver metastases.
* Adequate renal function: serum creatinine no more than 1.5 LSR or calculated creatinine clearance 60 ml / min (Crock).

Exclusion Criteria:

* The patient has received systemic cancer treatment within two weeks prior to extraction of the blood sample.
* Patient has received therapeutic radioisotopes such as strontium 89 within 4 weeks before blood extraction.
* Patient has had major surgery or percutaneous procedures such as placement of central venous catheter within 2 weeks prior to the blood draw.
* Patient has a history as bone marrow transplantation and / or stem cell transplantation.
* Patient has any of the following concomitant diseases or current conditions:

chronic active liver disease of any origin, and / or cirrhosis with Child-Pugh score B or C.

Uncontrolled active infection. carries the human immunodeficiency virus (HIV). Any other significant disease that in the opinion of the investigator, substantially increase the risk associated with patient participation in this study.

documented symptomatic brain metastases, progression or requiring corticosteroids or associated to a leptomeningeal involvement.

Patients with uncontrolled systemic diseases. Patients with Hypertension or Diabetes Mellitus is countable if at the time of inclusion deemed medically controlled.

Patients with inability for oral drug delivery, either by preventing gastrointestinal administration situation or severe impairment of intestinal absorption

* Any medical or psychiatric condition that, in the opinion of the investigator, may limit the patient's ability to understand and fulfill all requirements under its partcipación in the study.
* Pregnant or lactating women

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2012-11; Primary Completion 2012-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Overall survival | 12 months
  To determine the tumor progression-free survival at 3 and 6 months (PFS3 and PFS6) in both groups of patients and identify whether there is a statistically significant difference
gene expression profiles | 12 months
  Assess the correlation between the gene expression profiles obtained from the CTC and the gene expression profiles obtained from tumor samples from the same patients.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Gómez, M.D.,Ph.D, Study Director — Centro Nacional de Investigaciones Oncológicas (CNIO)
Locations (2):
- Spain (2):
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Madrid Norte Sanchinarro, Madrid, Madrid